CLINICAL TRIAL: NCT05002257
Title: Impact of Listening to Music on Anxiety Postoperative in a Postanesthesic Care Unit (PACU) After Spinal Anesthesia
Acronym: MusicAnx-SSPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PP21063
Record Dates: First submitted 2021-08-03; First posted 2021-08-12 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Spinal Anesthesia
Keywords: PACU; pain; care; music; anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental)
  Interventions: Other: music therapy
- Control arm (Active Comparator)
  Interventions: Other: No music therapy

INTERVENTIONS:
Other: music therapy — Patients included in the intervention arm with music therapy will choose among 3 possible music: music from elsewhere, classical music, today's music. These 3 music thearpy will have an identical duration of 20 minutes.
  Arms: Experimental Arm
Other: No music therapy — Usual care
  Arms: Control arm

SUMMARY:
Our hypothesis is that listening to music has a beneficial effect on the French population receiving spinal anesthesia for a scheduled procedure. We think we can reduce anxiety when switching to SSPI, using creative music therapy software (Music Care) French validated by clinical research.

DETAILED DESCRIPTION:
We want to demonstrate that listening to music:

* decreases the anxiety of patients in PHC;
* improves their overall satisfaction unlike patients subjected to ambient noise from the SSPI. Demonstrate that there is a link between trait anxiety assessed preoperatively and state anxiety assessed immediate postoperative period to anticipate and improve patient care as soon as they arrive in SSPI. Extend music listening to all patients staying in a postoperative SSPI or for procedures performed in SSPI (bladder probing, central venous approach, post locoregional analgesia operative…) The Music Care software that we have chosen to use has been specifically developed to use the music as a therapeutic aid. Numerous abstracts and clinical studies have been published on the subject the use of this software in reducing anxiety, pain, behavioral and changes in hemodynamic parameters. It is based on the use of the so-called "U" method, which is a relaxation method based on hypno-analgesia, thus offering a complete relaxation session to patient.

ELIGIBILITY:
inclusion criteria :

* adult patients;
* undergoing scheduled orthopedic surgery, under spinal anesthesia;
* non-cancerous, functional;
* in traditional or outpatient hospitalization;
* requiring a passage in PACU;
* agreeing to participate in the study (consent form).

exclusion criteria :

* Children;
* under tutorship or curatorship;
* having known hearing problems (hearing loss or not, deafness) reported during the anesthesia consultation or detected during the collection of preoperative data; having cognitive disorders (dementia, disorientation) reported during the consultation of anesthesia, not allowing questions to be answered
* Patients equipped with their personal music.

The following will be excluded when they arrive in SSPI:

* Patients who received a benzodiazepine during the intraoperative period;
* Patients whose spinal anesthesia has been converted to general anesthesia;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-07-08 (Actual)

PRIMARY OUTCOMES:
anxiety postoperative in a postanesthesic care unit (PACU) after spinal anesthesia | Day 0
  Anxiety is assess by using Spielberg's STAI-Ya from 20 (no anxiety) to 80 (anxiety)

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France